CLINICAL TRIAL: NCT05389904
Title: A Pre-emptive Prevention Bundle for Patients at High Risk for Hospital-onset Clostridioides Difficile
Brief Title: Pre-emptive Prevention for Patients at High Risk for Hospital-onset Clostridioides Difficile
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Pilgrim Health Care Institute (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); Massachusetts Host-Microbiome Center (Unknown); Hatch Family Foundation (Unknown)
Responsible Party: Principal Investigator, Meghan A. Baker, M.D, Associate Hospital Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022P000819
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: C. Difficile
Keywords: Prevention; Hospital-acquired infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients colonized with toxigenic C. difficile who do not receive the prevention bundle (Active Comparator): Patients colonized with toxigenic C. difficile, identified by testing routinely collected swabs for vancomycin-resistant enterococcus screening, who receive standard of care
  Interventions: Other: Arm 1: Routine care
- Patients colonized with toxigenic C. difficile who receive the prevention bundle (Active Comparator): Patients colonized with toxigenic C. difficile, identified by testing routinely collected swabs for vancomycin-resistant enterococcus screening, who receive a preemptive prevention bundle for C. difficile including enhanced room cleaning, C. difficile precautions, pharmacist review and optimization of antibiotics and antacids, and consideration of vancomycin prophylaxis.
  Interventions: Other: Arm 2: Preemptive C. difficile infection prevention bundle

INTERVENTIONS:
Other: Arm 1: Routine care — Patients colonized with toxigenic C. difficile, identified by testing routinely collected swabs for vancomycin-resistant enterococcus screening, will receive standard of care.
  Arms: Patients colonized with toxigenic C. difficile who do not receive the prevention bundle
Other: Arm 2: Preemptive C. difficile infection prevention bundle — Patients colonized with toxigenic C. difficile, identified by testing routinely collected swabs for vancomycin-resistant enterococcus screening, will receive a preemptive prevention bundle for C. difficile. The prevention bundle will include enhanced room cleaning, C. difficile precautions (staff entering room must wear gown and gloves and wash hands with soap and water upon exiting the room), pharmacist review and optimization of antibiotics and antacids, and consideration of vancomycin prophylaxis.
  Arms: Patients colonized with toxigenic C. difficile who receive the prevention bundle

SUMMARY:
Clostridioides difficile (C. difficile) is the most common healthcare-associated pathogen, causing >500,000 infections and >29,000 deaths per year in the US. Traditional approaches to reduce hospital-onset CDI focus on identifying, isolating, and treating symptomatic patients to prevent transmission to other patients. Recent genomic epidemiology studies, however, suggest that most hospital-onset CDI cases are attributable to asymptomatic carriers who either progress from colonization to active infection themselves or transmit C. difficile to other patients while asymptomatic. This trial will evaluate an intervention to pre-emptively identify asymptomatic C. difficile carriers and then implement a patient-tailored prevention package to protect the carrier from progression to active infection and to prevent transmission from the carrier to other patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU or Oncology units and identified to carry C. Difficile via VRE swab

Exclusion Criteria:

* Patients not identified as carriers of C. difficile and patients not admitted to ICU or oncology units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Risk of C. difficile infection among patients colonized with C. difficile comparing the intervention to the control group | 24 months
  Incidence rate ratio of CDI in colonized patients who received the intervention bundle versus who did not receive the intervention bundle

OTHER OUTCOMES:
Oncology and ICU C. difficile infection rates | 24 months
  Oncology and ICU C. difficile infection incidences before and after implementation of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Meghan A Baker, MD, SCD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No